CLINICAL TRIAL: NCT02493244
Title: Lipid Layer Thickness Pre and Post Lid Scrubs With Cliradex
Acronym: HONDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Canadian Optometric Education Trust Fund (COETF) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20714
Record Dates: First submitted 2015-06-08; First posted 2015-07-09 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants clean their eyelids with Cliradex wipes before going to bed at night.
  Interventions: Other: Cliradex
- Control (No Intervention): No treatment

INTERVENTIONS:
Other: Cliradex — Cliradex is simply water and 4-Terpineol, a natural organic compound found Melaleuca alternifolia. The other ingredients in Cliradex are in less than 1% of the formulation and are Glycerin, Polysorbate 20, Polysorbate 80, Carbomer, Triethanolamine.
  Arms: Treatment

SUMMARY:
Tears play a vital role in vision. A thin layer of tears is always present to cover the surface of the eye for optimal comfort and vision. There are several layers to the tear film, and the outer most layer is comprised of lipids. This lipid layer prevents evaporation of the tears and may be disrupted in people suffering from symptoms of dry eye. Cleaning eyelids with Cliradex wipes have shown to be effective in reducing dry eye symptoms in some patients, and the purpose of this study is to evaluate the tear film lipid layer thickness before and after one months treatment with Cliradex Wipes.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Have not worn contact lenses in the past month;
5. Has symptomatic dry eye with SPEED questionnaire score ≥6;
6. Corneal staining grade ≥2 on the Oxford scale.

Exclusion Criteria:

1. Has any known active ocular disease and/or infection;
2. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
3. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
4. Have used rewetting drops for a period of 2 days prior to screening visit;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment by verbal confirmation at the screening visit;
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Has taken part in another (pharmaceutical) research study within the last 30 days.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Lipid layer thickness | Baseline
  Lipid layer thickness measured in nm.
Lipid layer thickness | 1 month after baseline visit.
  Lipid layer thickness measured in nm.

SECONDARY OUTCOMES:
Non-invasive tear breakup time (NITBUT) | Baseline
  Measurement of time taken for a dry spot to appear on the corneal surface after blinking.
Non-invasive tear breakup time (NITBUT) | 1 month after baseline visit.
  Measurement of time taken for a dry spot to appear on the corneal surface after blinking.
Dry Eye Questionnaire (SPEED score) | Baseline
  Standard Patient Evaluation of Eye Dryness questionnaire. Assessment of subjects' frequency and severity of dry eye symptoms. The total score was calculated as the sum scores for all symptoms over a range of 0 to 28. A lower total SPEED score represents less frequent and/or less severe symptoms.
Dry Eye Questionnaire (SPEED score) | 15 days after baseline visit.
  Standard Patient Evaluation of Eye Dryness questionnaire. Assessment of subjects' frequency and severity of dry eye symptoms. The total score was calculated as the sum scores for all symptoms over a range of 0 to 28. A lower total SPEED score represents less frequent and/or less severe symptoms.
Dry Eye Questionnaire (SPEED score) | 1 month after baseline visit.
  Standard Patient Evaluation of Eye Dryness questionnaire. Assessment of subjects' frequency and severity of dry eye symptoms. The total score was calculated as the sum scores for all symptoms over a range of 0 to 28. A lower total SPEED score represents less frequent and/or less severe symptoms.
Overall corneal staining grade | Baseline
  Overall corneal staining score evaluated on a scale from 0 (none) to 5 (severe). A lower grade indicates less corneal surface desiccation.
Overall corneal staining grade | 1 month after baseline visit.
  Overall corneal staining score evaluated on a scale from 0 (none) to 5 (severe). A lower grade indicates less corneal surface desiccation.
Conjunctival hyperemia | Baseline
  Conjunctival hyperemia evaluated on a scale from 0 (negligible) to 100 (severe).
Conjunctival hyperemia | 1 month after baseline visit.
  Conjunctival hyperemia evaluated on a scale from 0 (negligible) to 100 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, Principal Investigator — CCLR, University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada